CLINICAL TRIAL: NCT04685811
Title: Evaluation of a 68Ga Small Molecule PSMA Antagonist Produced by Two Different Methods
Brief Title: Evaluation of PSMA Antagonist Produced by Two Different Methods
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-11021092; 7R01CA207645-03 (NIH)
Record Dates: First submitted 2020-12-02; First posted 2020-12-28 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Metastatic Prostate Adenocarcinoma
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 68Ga-PSMA-generator vs. 68Ga-PSMA-cyclotron (Experimental): Patients with metastatic prostate cancer will undergo two protocol 68Ga-PET scans within 24-48 hours with 68Ga-PSMA-cyclotron and 68Ga-PSMA-generator radiotracers.
  Interventions: Drug: 68Ga-PSMA-generator vs. 68Ga-PSMA-cyclotron

INTERVENTIONS:
Drug: 68Ga-PSMA-generator vs. 68Ga-PSMA-cyclotron — 68Ga-PSMA-generator vs. 68Ga-PSMA-cyclotron; single dose each, approximately 100-300 mBq.
  Other Names: Prostate specific membrane antigen imaging (PSMA)

SUMMARY:
Patients with metastatic prostate cancer will undergo two protocol 68Ga-PET scans within 24-48 hours with 68Ga-PSMA-cyclotron and 68Ga-PSMA-generator radiotracers. The goal of the study is to evaluate repeatability and equivalence across the different 68Ga-PSMA production methods. This research study is being conducted to assess whether the PET/CT imaging results, as generated from the two different 68Ga production methods, are equivalent.

DETAILED DESCRIPTION:
Patients with metastatic prostate adenocarcinoma will be enrolled in the study and will undergo two 68Ga-Prostate Specific Membrane Antigen- Positron Emission Tomography (PSMA-PET) scans within 24-48 hours. The difference between the two scans is that the radiotracer used in each scan will be produced with a different method (68Ga-PSMA-cyclotron and 68Ga-PSMA-generator produced). The first scan will occur after a baseline clinical evaluation, which will include a history, physical, and baseline lab draw. After each scan, blood draws will be obtained.

The purpose of this study is to evaluate equivalence of two processes to create 68Ga-HBED-PSMA and compare dosimetry, biodistribution and whole body excretion/ metabolism. Furthermore, the research team will perform dynamic analysis of the PET scans to investigate repeatability of whole-body 68Ga-PSMA-generator Ki Patlak imaging against that of conventional whole-body 68Ga-PSMA- SUV imaging and evaluate equivalence of whole-body 68Ga-PSMA Ki Patlak imaging between the two processes to create 68Ga-HBED-PSMA (68GA-PSMA-cyclotron vs. 68Ga-PSMA-generator). Patients will afterwards receive standard of care treatment and follow up imaging.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled in this study:

* Aged 21 years or older and below 80 years of age
* Signed written informed consent and willingness to comply with protocol requirements
* Histologically confirmed diagnosis of metastatic prostate cancer
* Staging imaging exam confirming metastatic disease, e.g. total body MRI, or CT chest/abdomen/pelvis, 99mTc bone scan, NaF PET

Exclusion Criteria:

* Laboratory values:
* Serum creatinine >2.5 mg/dL
* AST (SGOT) >2.5x ULN
* Bilirubin (total) >1.5x ULN
* Serum calcium >11 mg/dL
* Presence of any other co-existing condition which, in the judgment of the investigator, might increase the risk to the subject.
* Presence of serious systemic illness, including: uncontrolled inter-current infection, uncontrolled malignancy, significant renal disease, or psychiatric/social situations, which might limit compliance with study requirements.
* Other severe acute or chronic medical condition(s) or laboratory abnormality(ies) that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Inability to lay on the scanner table for the required period of time, e.g., due to bone pain or claustrophobia.

Ages: 21 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph R Osborne, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Generator PSMA Scan vs Cyclotron PSMA Scan: Intraclass Correation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax.
  Patients with metastatic prostate adenocarcinoma were administered a single intravenous dose approximately 100-300mBq of each of the study drugs 68Ga-PSMA-cyclotron and 68Ga-PSMA-generator 24- 48 hours apart.
  Intervention Description: 68Ga-PSMA-cyclotron and 68Ga-PSMA-generator; single dose each, approximately 100-300 mBq
Period: Overall Study
Arm/Group | Generator PSMA Scan vs Cyclotron PSMA Scan
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- ICC Between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax: Intraclass Correlation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax
Arm/Group | ICC Between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] — Subjects with a diagnosis of metastatic prostatic adenocarcinoma who meet the inclusion and exclusion criteria will be eligible for participation in this study. Therefore, baseline measures (age and sex) are collected prior to study enrollment.
  years | 73 [21 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Equivalence Between 68GA-PSMA-cyclotron and 68Ga-PSMA-generator Across Varying Pathologic Lesions
Description: Single score Intraclass Correlation Coefficient (ICC) was calculated as an index for reliability between 68GA-PSMA-cyclotron versus 68Ga-PSMA-generator across varying pathologic lesions. The ICC, based on a one-way random effects model was used to assess reliability. The ICC ratios in this data shows the top five lesions with the greatest PSMA uptake (SUV) in each patient. This is a measure of the variance of interest (for the patient's lesion) over the total variance (from all data points for that particular lesion of interest). Repeatability was evaluated by calculating the variance among group means of the SUVmean and SUVmax of each reference and lesion over the sum of the group-level and datalevel (residual) variance. The lesions reported in this analysis range from the SUV of reference organs to the average SUV of a metastatic deposit. These scans were also performed within 48 hours of each other to limit heterogeneity that may correspond to disease progression or PSMA avidity.
Time Frame: 2 study visits between 24 to 48 hours apart
Measure: Number (95% Confidence Interval); unit: ICC estimate
Groups:
- Comparison of Generator PSMA Scan vs. Cyclotron PSMA Scan: Intraclass Correlation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan
Arm/Group | Comparison of Generator PSMA Scan vs. Cyclotron PSMA Scan
Number analyzed (Participants) | 16
ICC estimate
  Lesion 1 | 0.98 [0.94 to 0.99]
  Lesion 2 | 0.98 [0.95 to 0.99]
  Lesion 3 | 0.99 [0.96 to 1.00]
  Lesion 4 | 0.99 [0.96 to 1.00]
  Lesion 5 | 0.97 [0.91 to 0.99]

2. Primary Outcome: Evaluate Equivalence Between 68GA-PSMA-cyclotron and 68Ga-PSMA-generator Across Varying Average SUV Max-pathologic Regions
Description: Single score intraclass correlation coefficient (ICC) was calculated as an index for reliability between 68GA-PSMA-cyclotron versus 68Ga-PSMA-generator across varying average SUV Max-pathologic regions
  The ICC ratios in this data provides a general performance review of uptake in both pathological lesions and reference lesions, specifically the average SUVmax of bone metastases, lymph nodes, salivary glands, and the spleen.
Time Frame: 2 study visits between 24 to 48 hours apart
Measure: Number (95% Confidence Interval); unit: ICC estimate
Groups:
- Comparison of Generator PSMA Scan vs Cyclotron PSMA Scan: Intraclass Correlation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan: Average SUV Max
Arm/Group | Comparison of Generator PSMA Scan vs Cyclotron PSMA Scan
Number analyzed (Participants) | 16
ICC estimate
  Average SUV Max - Bone Lesions | 0.96 [0.88 to 0.99]
  Average SUV Max - Lymph Nodes | 0.86 [0.62 to 0.95]
  Average SUV Max - Salivary Glands and Parotids | 0.70 [0.34 to 0.88]
  Average SUV Max - Spleen | 0.82 [0.57 to 0.93]

3. Primary Outcome: ICC Between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax
Description: Repeatability was evaluated by calculating the variance among group means of the SUVmean and SUVmax of each reference and lesion over the sum of the group-level and datalevel (residual) variance. The intraclass correlation coefficient (ICC), based on a one-way random effects model (i.e., assumes subjects are randomly selected from the larger population), was used to assess reliability between generator and cyclotron scanning methods. BlandAltman analysis evaluated the agreement between the two scanning methods. Confidence levels of 95% were estimated to assess precision of the obtained estimates. All analyses were performed in R Version 4.0.5 (R Foundation for Statistical Computing, Vienna, Austria).
Time Frame: 2 study visits between 24 to 48 hours apart
Measure: Number; unit: ICC estimate
Arm/Group | ICC Between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax
Number analyzed (Participants) | 16
ICC estimate | 0.97

4. Secondary Outcome: Evaluate Equivalence Between 68GA-PSMA-cyclotron and 68Ga-PSMA-generator Across Varying Max SUV -Pathologic Regions
Description: Single score intraclass correlation coefficient (ICC) was calculated as an index for reliability between 68GA-PSMA-cyclotron versus 68Ga-PSMA-generator across varying Max SUV -pathologic regions
  Repeatability was evaluated by calculating the variance among group means of the SUVmean and SUVmax of each reference and lesion over the sum of the group-level and datalevel (residual) variance. The intraclass correlation coefficient (ICC), based on a one-way random effects model (i.e., assumes subjects are randomly selected from the larger population), was used to assess reliability between generator and cyclotron scanning methods. BlandAltman analysis evaluated the agreement between the two scanning methods. Confidence levels of 95% were estimated to assess precision of the obtained estimates. All analyses were performed in R Version 4.0.5 (R Foundation for Statistical Computing, Vienna, Austria).
Time Frame: 2 study visits between 24 to 48 hours apart
Measure: Number (95% Confidence Interval); unit: ICC estimate
Groups:
- Comparison of Generator PSMA Scan vs Cyclotron PSMA Scan: MAX SUV: Intraclass Correlation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan: MAX SUV
Arm/Group | Comparison of Generator PSMA Scan vs Cyclotron PSMA Scan: MAX SUV
Number analyzed (Participants) | 16
ICC estimate
  Max SUV - Aorta | 0.59 [0.17 to 0.84]
  Max SUV - Liver | 0.91 [0.76 to 0.97]
  Max SUV - Parotid | 0.78 [0.48 to 0.92]

5. Secondary Outcome: Compare Bio-Distribution Between 68GA-PSMA-cyclotron vs. 68Ga-PSMA-generator
Description: The biodistribution of 68GA-PSMA-cyclotron versus 68Ga-PSMA-generator will be evaluated by measuring the radioactivity concentration in various organs of interest. Based on the SUVmean and SUVmax, the RC unit will be used to compare these scans.
  PSMA positivity was defined as having a SUV value above that of the reference blood pool, liver, and/or salivary glands when evaluating lesions as described using the PROMISE criteria15. Quantitative analysis reviewed the SUVmax and SUVmean of the parotid gland, liver, and aortic arch (blood pool), as well as the SUVmax and SUVmean of suspected metastatic lesions. The same ROIs were evaluated on both scans for each respective patients.
Time Frame: 2 study visits between 24 to 48 hours apart
Measure: Number (95% Confidence Interval); unit: ICC estimate
Groups:
- Comparison Between Generator PSMA vs Cyclotron PSMA: Intraclass Correlation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan
Arm/Group | Comparison Between Generator PSMA vs Cyclotron PSMA
Number analyzed (Participants) | 16
ICC estimate
  Total Lesion Average Coefficient Variation | 0.97 [0.92 to 0.99]
  Total Lesion Average Standard Deviation | 0.94 [0.85 to 0.98]
  Total Lesion Average SUV Max | 0.97 [0.91 to 0.99]
  Total Lesion Average SUV Mean | 0.71 [0.36 to 0.89]

ADVERSE EVENTS:
Time Frame: Each participant will have adverse events data collected at each study visit (2 visits total). At each study visit, the investigator will inquire about the occurrence of AE/SAEs since the last visit.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 will be utilized for AE reporting.
  HBED-PSMA has been injected for PET imaging in more than 500 published patients. No drug related side effects have been observed. This is expected because the mass of compound is minimal, less than 10 micrograms.
Groups:
- Generator PSMA Scan vs Cyclotron PSMA Scan: Intraclass Correlation Coefficient (ICC) between Generator PSMA Scan vs Cyclotron PSMA Scan: Total Lesion Average SUVMax
Arm/Group | Generator PSMA Scan vs Cyclotron PSMA Scan
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
The small sample size which resulted from recruitment and logistical challenges was a limiting factor in the analytical interpretation. It is important to note that the purpose of the study was to determine if the equivalency can also translate to mass production in the clinical setting. Future studies should evaluate the cost-benefit analysis of 68Ga based radioisotopes with 18F. We anticipate that production of 68GaPSMA cyclotron is a cost-efficient method of 68Ga production for clinical use.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/11/NCT04685811/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/11/NCT04685811/ICF_001.pdf